CLINICAL TRIAL: NCT04292808
Title: An Open-Label Study to Assess the Efficacy and Safety of Low Dose Methoxyflurane (PENTHROX®) for Pain Control During Outpatient Aesthetic Surgeries and Facial Filler Injections
Brief Title: Low Dose Methoxyflurane and Out-Patient Aesthetic Surgery and Facial Filler
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid caused too many delays
Sponsor: Verso Surgery Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: PRO00040577
Record Dates: First submitted 2020-02-27; First posted 2020-03-03 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Methoxyflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Penthrox (Other): Low Dose Methoxyflurane
  Interventions: Drug: Methoxyflurane

INTERVENTIONS:
Drug: Methoxyflurane — Methoxyflurane inhaler during out-patient aesthetics surgery or facial dermal fillers.
  Other Names: Penthrox

SUMMARY:
The aim of the study is to generate real-world evidence on the effectiveness, safety and additional parameters of low dose methoxyflurane (PENTHROX®) in: aesthetic surgeries (eg. hair transplant, upper blepharoplasty, otoplasty, upper brow lift, and mentoplasty) and facial filler injections [eg. hyaluronic acid (HA) and Sculptra®] in an outpatient aesthetic practice. This will be an open-label study, with a total of 60 patients undergoing a planned outpatient aesthetic surgery or filler injection (30 patients in each group).

ELIGIBILITY:
Inclusion Criteria:

1. Conscious adult patients: ≥ 18 years of age
2. Patient is scheduled for an outpatient anesthetic surgery (eg. hair transplant, upper blepharoplasty, otoplasty, upper brow lift, and mentoplasty) or a facial filler injection (eg. HA, and Sculptra®).
3. Patient should understand the nature of the study and provide written informed consent
4. Patient is able to follow all study requirements and procedures and complete required questionnaires

Exclusion Criteria:

1. An altered level of consciousness, due to any cause, including head injury, drugs, or alcohol
2. Clinically significant renal impairment
3. Women of child bearing potential who are pregnant or peri partum, including labour
4. A history of liver dysfunction after previous methoxyflurane use or other halogenated anesthetics
5. Hypersensitivity to methoxyflurane or other halogenated anesthetics, or to butylated hydroxytoluene
6. Known or genetically susceptible to malignant hyperthermia or a history of severe adverse reactions in either patient or relatives
7. Clinically evident or potential hemodynamic instability as per the opinion of the investigator
8. Clinically evident respiratory impairment as per the opinion of the investigator
9. Prior treatment with PENTHROX® within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Assessing patient satisfaction | through study completion, an average of 1 year
  Global assessment of medication performance (gmp)

CONTACTS AND LOCATIONS:
Locations (1):
- Verso Surgery Centre, Oakville, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Romagnoli A, Busque L, Power DJ. The "analgizer" in a general hospital: a preliminary report. Can Anaesth Soc J. 1970 May;17(3):275-8. doi: 10.1007/BF03004607. No abstract available. PMID 5512851
- See also: Penthrox Data Sheet - New Zealand (2017) — http://www.medsafe.govt.nz/profs/datasheet/p/penthroxinh.pdf